CLINICAL TRIAL: NCT05746975
Title: Diabetic Retinopathy Classification: ETDRS 7-fields vs Widefield Imaging (Clarus 500 and Optos California)
Brief Title: Diabetic Retinopathy Classification: ETDRS 7-fields vs Widefield Imaging (ClarusDR)
Acronym: ClarusDR
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Other Study IDs: 4C-2023-12
Record Dates: First submitted 2023-02-06; First posted 2023-02-28 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Retinopathy, Diabetic
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to analyse and compare Diabetic Retinopathy severity level using 30º ETDRS 7-fields and Wide-field Imaging techniques using Clarus 500 (Carl Zeiss Meditech Inc., Dublin, USA) and Optos (Optos, Dunfermline, UK) in diabetic patients with mild to moderate diabetic retinopathy. The main questions it aims to answer are:

1. To compare the Clarus 500TM wide-field imaging technique with the ETDRS 7-fields method in the assessment of DR severity level using the ETDRS DRSS.2. To compare the two wide-field imaging techniques (Clarus 500TM vs OptosTM) in the assessment of DR severity level using the ETDRS DRSS.3. To evaluate the peripheral area imaged by the wide-field Clarus 500TM and OptosTM to characterize DR lesions distribution (predominantly observed within or outside the ETDRS 7-fields) and severity (according to the ETDRS standard photos).4. To determine the relevance and frequency of DR PPL, located outside the ETDRS 7-fields area, and to explore PPL occurrence in different DR severity levels.

Participants will undergo a non-invasive ophthalmological examination, which includes BCVA, 7-fields CFP and UWF FP to assess ETDRS DRSS level.

DETAILED DESCRIPTION:
Diabetic Retinopathy (DR) remains a significant cause of blindness in working-age populations across the world. The gold-standard method for assessing its severity is the modified Airlie House classification developed for the Early Treatment Diabetic Retinopathy Study (ETDRS), still used by clinical trials for developing of DR therapeutic and management guidelines.

ETDRS Diabetic Retinopathy Severity Score (DRSS) is based on the identification of DR lesions on colour fundus photography's (CFP) obtained in different locations of the retina. The photography acquisition protocol consists in acquiring seven stereoscopic pairs of overlapping 30° fields images of the ocular fundus to map out the macula and mid-peripheral retina. Photographers and fundus camera systems usually need training and certification by external reading centres to guarantee proper images quality and fields definition in a process that can be challenging with a considerable learning curve. Patient collaboration to follow a fixation point in different locations and withstand intense flashes of light, a good dilation of eye pupil and the difficulty to obtain well focused images in peripherical gaze positions are some of the main difficulties for obtaining gradable images using this 7-fields acquisition protocol.

On the other side, the grading process of ETDRS 7-fields images can be extremely labour-intensive and strongly dependent on the quality of the images, presence of artifacts and the definition of the peripherical fields, requiring well-trained people to identify and recognise features that can be very subtle or easily get unnoticed.

Moreover, the retinal area documented with the ETDRS 7-fields protocol represents approximately only 35% of the retina surface. Substantial diabetic retinal pathology can exist in the retinal periphery located outside this area which is being emphasized by advanced retinal imaging technology. Predominantly Peripheral Lesions (PPL) like the presence of venous beading, new-vessels, haemorrhages and microaneurysms in the extreme periphery have been correlated with peripheral non-perfusion, neurodegenerative changes and consequent increase of DR progression.

Recent instrumentation like OptosTM (Optos, Dunfermline, UK) or Clarus 500TM (Carl Zeiss Meditech Inc., Dublin, USA) allow wide-field acquisitions that document up to 90% of the retina surface in just one or two images decreasing patients tiredness and discomfort and overcoming most of the quality and fields definition issues described above.

OptosTM equipment can acquire almost 200º of the retina in just one picture without the need for pupil dilation and using ultra-widefield scanning laser ophthalmoscopy (SLO) technology. Its final image is based on the superimposition of two images acquired with 2 different laser wavelengths: a green and a red wavelength, giving a semirealistic colour image that despite its high contrast and sharpness, gives the retina a greenish and unreal aspect. Also, its 200º field amplitude is usually disturbed by artifacts caused by the presence of eyelashes or eyelids, that mainly obscure the peripherical area of the retina.

On the other hand, Clarus 500 TM equipment uses an imaging technique called Broad Line Fundus Imaging that is a hybrid of confocal SLO (cSLO) and traditional fundus photography. This technology provides higher resolution images with more accurate coloration of the fundus. A single image capture with this system obtains 133-degrees of view but with the acquisition of just two pictures (a temporal and nasal image of the retina), a 200-degree of view can be achieved.

Several studies have suggested moderate to substantial agreement between Optos ultra-wide field (UWF) and ETDRS 7-fields imaging and have shown that DR occurs in areas peripheral to the ETDRS fields in up to 40% of eyes, which may imply a more severe level of DR in 9% to 15% of eyes. However, there is only limited data regarding the validity of DR assessment using Clarus 500TM imagine technique obtained in cross-sectional studies with few patients.

On this basis, the aim of this work is to identify and compare the ETDRS severity level of diabetic patients using 3 different images modalities: the 30º ETDRS 7-fields colour fundus photography's protocol, the 2 wide-field images technique with Clarus 500 TM and the 1 wide-field image of OptosTM, in a prospective, longitudinal, and randomized study. The ETDRS 7-fields area will be superimposed on both wide-field equipment's images so equivalent retinal areas will be analysed. Our goal is to demonstrate that ETDRS severity level can be accurately evaluated using only two Clarus 500TM high quality images with wider amplitude, decreasing the effort and collaboration skills that are required in older techniques, while improving the quality and identification capability of key disease features with less artifacts than other wide-field systems. Additionally, peripheral retina outside the ETDRS 7-fields area will also be analysed to assess the presence of PPL and evaluate its relevance and association with disease severity level and progression.

Finally, the investigators expect to evaluate patients' opinion about their experience in each imaging modality, evaluating their discomfort and satisfaction degree while submitted to each procedure.

ELIGIBILITY:
Inclusion Criteria:

* DM type 2 according to 1985 World Health Organization (WHO) criteria
* Age between 35 and 80 years
* BCVA ≥ 75 letters (20 /32)
* Refraction with a spherical equivalent less than 5 Diopters
* NPDR levels 35 and 43-47 (based on the ETDRS criteria - 7 fields CFP)

Exclusion Criteria:

* Cataract or other eye disease that may interfere with fundus examinations
* Glaucoma
* Other retinal vascular disease than DR
* Refractive errors > to + or - 5 Diopters
* Pupil diameter of less than 5 mm
* Poor quality images due to artifacts, movements, or media opacities

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic type 2 patients with mild to moderate/severe NPDR
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
ETDRS severity level according to the Early Treatment Diabetic Retinopathy Study - Diabetic Retinopathy Severity Scale (ETDRS-DRSS). | 12 months
  Compare DR severity level between the ETDRS 7-fields imaging and the wide-field imaging techniques: Clarus 500TM and OptosTM. The ETDRS - DRSS goes from level 10 - no presence of DR to level 75 - Severe proliferative DR
One or more than 2-steps change on ETDRS - DRSS severity level | 12 months
  Compare ETDRS -DRSS between the two imaging techniques and evaluate the presence of 1 step or more than 2 steps difference between ETDRS 7-fields imaging and the wide-field imaging techniques: Clarus 500TM and OptosTM
Peripheral DR lesions characterization | 12 months
  Investigate the peripheral area and analyze the presence, distribution, and severity of peripheral DR lesions, in wide-field images: Clarus 500TM and OptosTM.
  Presence and distribution of lesions in the periphery will be evaluated as 1) Not observed; 2) predominantly observed outside ETDRS fields; 3) Uniformly distributed within and outside ETDRS fields. 4) Ungradable.
  Severity of the peripheral lesions will be evaluated using the same ETDRS-DRSS scale described above and will vary between level 35 and level 65.
  Also, it will then be compared with the ETDRS 7-field area and graded as less, equivalent or greater than the observed inside ETDRS 7-fields area.

SECONDARY OUTCOMES:
Evaluation of Images quality in each imaging modality. | 12 months
  Images from each modality (7-fields, Clarus 500 and Optos TM) will be analysed according to 1) presence of artifacts like eyelashes, halos, eyelids, cataract opacities, etc; 2) Presence of unfocused areas 3) % of area occupied by those artifacts.
Evaluation of Patients satisfaction about each imagining modality. | 12 months
  To evaluate patient's experience and degree of satisfaction in each imaging modality, a questionnaire will be developed with qualitative and quantitative questions covering all aspects of the experience.
Correlate and analysed DR findings in each imaging technique with disease severity | 12 months
  To characterize the study population, demographic, and systemic characteristics, as well as visual function (BCVA), will be collected and analysed to correlate DR findings in each imaging technique with disease severity

CONTACTS AND LOCATIONS:
Overall Officials: Ana R Santos, PhD, Principal Investigator — Association for Innovation and Biomedical Research on Light and Image
Locations (1):
- AIBILI-CEC (AIBILI- Clinical Trials Centre), Coimbra, Portugal

REFERENCES:
- [Background] Shimizu K, Kobayashi Y, Muraoka K. Midperipheral fundus involvement in diabetic retinopathy. Ophthalmology. 1981 Jul;88(7):601-12. doi: 10.1016/s0161-6420(81)34983-5. PMID 6167923
- [Background] Wessel MM, Aaker GD, Parlitsis G, Cho M, D'Amico DJ, Kiss S. Ultra-wide-field angiography improves the detection and classification of diabetic retinopathy. Retina. 2012 Apr;32(4):785-91. doi: 10.1097/IAE.0b013e3182278b64. PMID 22080911
- [Background] Silva PS, Cavallerano JD, Haddad NM, Kwak H, Dyer KH, Omar AF, Shikari H, Aiello LM, Sun JK, Aiello LP. Peripheral Lesions Identified on Ultrawide Field Imaging Predict Increased Risk of Diabetic Retinopathy Progression over 4 Years. Ophthalmology. 2015 May;122(5):949-56. doi: 10.1016/j.ophtha.2015.01.008. Epub 2015 Feb 19. PMID 25704318
- [Background] Silva PS, Cavallerano JD, Sun JK, Soliman AZ, Aiello LM, Aiello LP. Peripheral lesions identified by mydriatic ultrawide field imaging: distribution and potential impact on diabetic retinopathy severity. Ophthalmology. 2013 Dec;120(12):2587-2595. doi: 10.1016/j.ophtha.2013.05.004. Epub 2013 Jun 15. PMID 23778092
- [Background] Chen A, Dang S, Chung MM, Ramchandran RS, Bessette AP, DiLoreto DA, Kleinman DM, Sridhar J, Wykoff CC, Kuriyan AE. Quantitative Comparison of Fundus Images by 2 Ultra-Widefield Fundus Cameras. Ophthalmol Retina. 2021 May;5(5):450-457. doi: 10.1016/j.oret.2020.08.017. Epub 2020 Aug 29. PMID 32866664
- [Background] Rasmussen ML, Broe R, Frydkjaer-Olsen U, Olsen BS, Mortensen HB, Peto T, Grauslund J. Comparison between Early Treatment Diabetic Retinopathy Study 7-field retinal photos and non-mydriatic, mydriatic and mydriatic steered widefield scanning laser ophthalmoscopy for assessment of diabetic retinopathy. J Diabetes Complications. 2015 Jan-Feb;29(1):99-104. doi: 10.1016/j.jdiacomp.2014.08.009. Epub 2014 Aug 28. PMID 25240716
- [Background] Silva PS, Cavallerano JD, Sun JK, Noble J, Aiello LM, Aiello LP. Nonmydriatic ultrawide field retinal imaging compared with dilated standard 7-field 35-mm photography and retinal specialist examination for evaluation of diabetic retinopathy. Am J Ophthalmol. 2012 Sep;154(3):549-559.e2. doi: 10.1016/j.ajo.2012.03.019. Epub 2012 May 23. PMID 22626617
- [Background] Wessel MM, Nair N, Aaker GD, Ehrlich JR, D'Amico DJ, Kiss S. Peripheral retinal ischaemia, as evaluated by ultra-widefield fluorescein angiography, is associated with diabetic macular oedema. Br J Ophthalmol. 2012 May;96(5):694-8. doi: 10.1136/bjophthalmol-2011-300774. Epub 2012 Mar 15. PMID 22423055
- [Background] Price LD, Au S, Chong NV. Optomap ultrawide field imaging identifies additional retinal abnormalities in patients with diabetic retinopathy. Clin Ophthalmol. 2015 Mar 24;9:527-31. doi: 10.2147/OPTH.S79448. eCollection 2015. PMID 25848202
- [Background] Matsui Y, Ichio A, Sugawara A, Uchiyama E, Suimon H, Matsubara H, Sugimoto M, Ikesugi K, Kondo M. Comparisons of Effective Fields of Two Ultra-Widefield Ophthalmoscopes, Optos 200Tx and Clarus 500. Biomed Res Int. 2019 Dec 5;2019:7436293. doi: 10.1155/2019/7436293. eCollection 2019. PMID 31886247
- [Background] Hirano T, Imai A, Kasamatsu H, Kakihara S, Toriyama Y, Murata T. Assessment of diabetic retinopathy using two ultra-wide-field fundus imaging systems, the Clarus(R) and Optos systems. BMC Ophthalmol. 2018 Dec 20;18(1):332. doi: 10.1186/s12886-018-1011-z. PMID 30572870
- [Background] Aiello LP, Odia I, Glassman AR, Melia M, Jampol LM, Bressler NM, Kiss S, Silva PS, Wykoff CC, Sun JK; Diabetic Retinopathy Clinical Research Network. Comparison of Early Treatment Diabetic Retinopathy Study Standard 7-Field Imaging With Ultrawide-Field Imaging for Determining Severity of Diabetic Retinopathy. JAMA Ophthalmol. 2019 Jan 1;137(1):65-73. doi: 10.1001/jamaophthalmol.2018.4982. PMID 30347105
- [Background] Grading diabetic retinopathy from stereoscopic color fundus photographs--an extension of the modified Airlie House classification. ETDRS report number 10. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1991 May;98(5 Suppl):786-806. PMID 2062513
- [Background] International Conference on Harmonisation of technical requirements for registration of pharmaceuticals for human use.. ICH harmonized tripartite guideline: Guideline for Good Clinical Practice. J Postgrad Med. 2001 Jan-Mar;47(1):45-50. No abstract available. PMID 11590294
- [Background] World Medical Association.. World Medical Association Declaration of Helsinki. Ethical principles for medical research involving human subjects. Bull World Health Organ. 2001;79(4):373-4. Epub 2003 Jul 2. No abstract available. PMID 11357217
- [Background] Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016 on the Protection of Natural Persons with Regard to the Processing of Personal Data and on the Free Movement of Such Data. Off. J. Eur. Union 2016, L119, 1-88; DOI: L:2016:119:TOC.